CLINICAL TRIAL: NCT00489749
Title: The Influence of Protected Early Weightbearing Versus Nonweightbearing After Surgical Repair of the Achilles Tendon
Brief Title: A Study Comparing Protected Early Weightbearing Versus Non-Weightbearing After Surgery for Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other); Edmonton Orthopaedic Research Society (Unknown); DonJoy Orthotics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JomhaAchillesEdm1
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; Open surgical repair; Early functional mobilization; Weightbearing; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Protected early weightbearing/Achilles tendon surgery

SUMMARY:
The purpose of this study was to determine the effect of protected early weightbearing (PEWB) compared to non-weightbearing (NWB) after surgery for an Achilles tendon rupture (ATR) on health related quality of life (HRQL) in the initial six week period after surgery, functional recovery over time, return to work and activity and complications. We hypothesized that PEWB following ATR repair would result in: i) improved HRQL in the initial postoperative period, ii), a quicker recovery of HRQL, strength and endurance, iii) earlier return to work and sport, and iv) no increase in complications, such as re-rupture compared to NWB.

DETAILED DESCRIPTION:
Achilles tendon rupture (ATR) is commonly treated with open surgical repair. Following surgical repair, there are a variety of protocols, ranging from complete immobilization to immediate postoperative mobilization with early weightbearing. However, no clear consensus regarding the optimal postoperative rehabilitation protocol for ATRs exists. Early rehabilitation after ATR has been shown to be beneficial in animal and human studies. Human prospective studies and randomized controlled trials have shown that early postoperative mobilization do not pose additional risks compared to cast immobilization, with a trend toward a reduction in lost work days and an earlier return to sport. However, these trials define early postoperative mobilization differently (i.e. use different combinations of weightbearing and range of motion). This makes it difficult to determine which factor in the early rehabilitation process plays an important role in optimizing recovery. An important component of early rehabilitation is weightbearing.

Comparison: Patients weightbearing in the early rehabilitation period after surgical repair of the Achilles tendon compared to patients non-weightbearing after the surgical repair of the Achilles tendon repair. With the exception of weightbearing status, both groups performed the same rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* closed and complete Achilles tendon rupture
* seen within 14 days of injury in hospital

Exclusion Criteria:

* unwilling to follow the study's rehabilitation protocol
* unable to speak or read English
* co-morbid conditions such as diabetes and neurological or collagen disease
* pregnancy
* recent immunosuppressant or fluoroquinolone therapy
* previous Achilles tendon symptoms
* previous ipsilateral rupture
* sustained an additional injury not allowing weightbearing
* an Achilles tendon avulsion injury
* unfit for surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Health related quality of life: Short form 36 questionnaire | six weeks

SECONDARY OUTCOMES:
Health related quality of life: Short Form-36 questionnaire | 3 and 6 months
Level of activity: tailored question | six weeks, 3 months, and 6 months
Major complications: chart review | 6 weeks, 3 months, and 6 months
Minor complications: chart review | 6 weeks, 3 months, and 6 months
Isometric muscle strength: hand held myometer | 6 weeks, 3 months, and 6 months
Muscle endurance: heel raise counting device | 6 months
Calf circumference: standardized tape measurement | 6 weeks, 3 months, and 6 months
Return to work/sport: tailored question | 6 weeks, 3 months, and 6 months
Physiotherapy utilization: tailored question | 6 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadr Jomha, MD, PhD, Principal Investigator — University of Alberta Division of Orthopaedic Surgery; Amar Suchak, MD, Study Director — University of Alberta Department of Medicine and Dentistry
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada